CLINICAL TRIAL: NCT00619229
Title: Confirmatory, Prospective, Randomized, Double-blind, Placebo-controlled, Parallel Groups Study to Assess the Efficacy and Safety of Prostaglandin E1 in Subjects With Dry Age-related Macular Degeneration.
Brief Title: Alprostadil in Maculopathy Study (AIMS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim Analysis: Optimization of study design required.
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0878; 2005-005686-11 (EudraCT Number)
Record Dates: First submitted 2007-12-24; First posted 2008-02-20 (Estimated); Results first posted 2011-04-11 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2011-11

CONDITIONS: Macular Degeneration
Keywords: Alprostadil; prostaglandin E1; Prostavasin®; macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Alprostadil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alprostadil (Experimental): Alprostadil
  Interventions: Drug: Alprostadil (prostaglandin E1)
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alprostadil (prostaglandin E1) — Alprostadil 20 µg ampoules; 60 µg alprostadil/d i.v. for 15 days.
  Other Names: Prostavasin
  Arms: Alprostadil
Other: Placebo — Placebo/d i.v. for 15 days
  Arms: Placebo

SUMMARY:
Evaluation of efficacy of alprostadil (prostaglandin E1) for treatment of patients suffering from dry age-related macula degeneration

DETAILED DESCRIPTION:
Results of the planned interim analysis indicated that the number of originally planned patients were not sufficient to reach statistical significance in the primary end point. Instead of increasing the sample size accordingly, it was decided to terminate the study and plan future proceedings based on a careful analysis of the unblinded results.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects older than 50 years of age.
* Dry age-related macula degeneration (AMD) with hard drusen and possibly beginning geographic atrophy in one eye
* Visual acuity between 0.2 and 0.7 (logMAR) assessed with ETDRS charts

Exclusion Criteria:

* Dry AMD AREDS category 3 or 4 in both eyes
* Wet AMD in at least one eye
* Detachment of the pigmentary epithelium
* Glaucoma
* Diabetic retinopathy
* Medical history of retinal vein occlusion
* Uveitis
* Cataract surgery during the study
* High myopia (< -6 dpt) with pathological findings of the retina
* Medical history of any opthalmic surgery with complications
* Medical history of cataract surgery without complications within the last 12 weeks
* Medical history of vitrectomy
* AREDS medication within the last 2 days
* Opthalmologic dietary supplements within the last 2 days
* Medical history of retinal hemorrhage
* Cardiac failure (NYHA grade II or higher)
* Inadequately controlled coronary heart disease or cardiac arrhythmia
* Subject has a medical history and/or suspicion of pulmonary edema or pulmonary infiltration
* Subject has a peripheral edema
* Myocardial infarction within 6 months prior to enrollment
* Subject has renal insufficiency, compensated retention (creatinine > 1,5 mg/dL)
* Subject has known existing malignant disease
* Severe chronic obstructive pulmonary disease
* Subject has a venoocclusive lung disease
* Known hepatic disease
* Inadequately controlled or untreated hypertension (systolic blood pressure ≥ 180 mmHg, diastolic blood pressure ≥ 110 mmHg)
* Subject has upper grade cardiac valvular disorders
* Pregnancy or lactation period
* Known hypersensitivity to PGE1 or to any component of the trial medication
* Subject has a history of chronic alcohol or drug abuse within the past 2 years
* Subject has known lactose intolerance
* Poor general state of health or other criteria
* Subject has other serious illness
* Laboratory values outside the normal range unless considered not clinically relevant by the investigator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (6):
- Germany (6):
  - Berlin
  - Bochum
  - Dortmund
  - Karlsruhe
  - München
  - Münster

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Product Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2011/021726s008lbl.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Full Analysis Set (FAS) includes all randomized subjects treated with at least one infusion and having valid Baseline and Post-Baseline measurements.
  The Randomized Set (RS) consists of all randomized subjects who have completed Visit 16 or terminated prematurely.
Pre-assignment Details: Participant Flow shows the RS. Baseline Characteristics refer to the FAS.
Groups:
- Alprostadil: Alprostadil 60 mcg/day i.v. for 15 days
- Placebo: Placebo i.v. for 15 days
Period: Overall Study
Arm/Group | Alprostadil | Placebo
Started | 18 | 18
Full Analysis Set (FAS) | 16 | 17
Completed | 14 | 16
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Termination of the Study by the Sponsor | 1 | 1
Not completed — Investigator planned Cataract Operation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alprostadil | Placebo | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (8.5) | 71.7 (8.1) | 73.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 10 | 8 | 18
White [Number; unit: participants] | 16 | 17 | 33
Weight [Mean (Standard Deviation); unit: kilogramm (kg)] | 77.14 (14.71) | 76.46 (14.49) | 76.79 (14.37)
Height (cm) [Mean (Standard Deviation); unit: centimeter (cm)] | 171.06 (9.29) | 168.59 (8.69) | 169.79 (8.93)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/ (m^2)] | 26.20 (3.38) | 26.70 (3.32) | 26.45 (3.31)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Visual Acuity Between Measurements at 3 Months After Drug Intervention and Measurements at Baseline (Assessed Within Early Treatment Diabetic Retinopathy Study (ETDRS) Chart)
Description: Difference in visual acuity was measured with the standard ETDRS chart with letters arranged in lines of five. The first line is assumed to have letters of a specific size and each subsequent line to consist of letters of a smaller size. The subject starts reading the first line and continues reading the following lines until failing a line. Passing a line means to name at least three of the five letters correctly.
Time Frame: From baseline to 3 months
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Lines read in ETDRS chart
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Lines read in ETDRS chart | 0.94 (1.84) | 0.53 (1.66)
Statistical Analysis 1: Comparison: Alprostadil vs Placebo; The primary goal of the study was to test the following null hypothesis: H0: μAlprostadil ≤ μPlacebo, against the alternative hypothesis H1: μAlprostadil > μPlacebo, where μ denotes the mean differences in visual acuity between measurements at 3 months after the end of study drug infusion minus measurements at baseline as assessed as line difference on the standard ETDRS charts; Test type: Superiority or Other; p = 0.1220, ANCOVA — The criterion for significance (α) was set at one-sided α = 0.025, which means that only an effect in the expected direction was interpreted; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [-0.674 to 2.55] — For exploratory testing an Analysis of Variance-Covariance (ANCOVA) F-test with dependent variable 'difference in visual acuity', fixed factors 'treatment' and 'centre' and Baseline value as a covariate was used

2. Secondary Outcome: The Difference in Visual Acuity Between Measurements Immediately After Intervention and Measurements at Baseline
Description: as for outcome 1
Time Frame: From baseline to time immediately after intervention
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Lines read in ETDRS chart
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Lines read in ETDRS chart | 1.29 (1.44) | 0.38 (1.54)

3. Secondary Outcome: The Difference in Visual Acuity Between Measurements at 6 Months After Intervention and Measurements at Baseline
Description: as for outcome 1
Time Frame: From baseline to 6 months
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Lines read in ETDRS chart
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Lines read in ETDRS chart | 1.31 (1.45) | 0.29 (2.11)

4. Secondary Outcome: Progression of the Dry Age-related Macular Degeneration
Description: Severity of the diagnosed dry age-related macular degeneration (AMD) was assessed in comparison to Baseline and classified as
  1. Progression
  2. Stabilization
  3. Amelioration
Time Frame: From baseline to 6 months
Population: Full Analysis Set (FAS)
Measure: Number; unit: Participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Participants
  Progression in disease | 11 | 10
  Stabilization of disease | 1 | 3
  Amelioration of disease | 4 | 4

5. Secondary Outcome: Development of a Wet Age-related Macular Degeneration
Description: A wet age-related macular degeneration (AMD) is defined as the development of choroidal neovascularization of the "study-eye" (worse eye).
  Development is categorized in Yes and No, where Yes means that a subject who had no wet AMD at Screening has developed a wet AMD at Week 29.
Time Frame: From baseline to 6 months
Population: Full Analysis Set (FAS)
Measure: Number; unit: Participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Participants
  Yes | 0 | 0
  No | 16 | 17

6. Secondary Outcome: The Difference in Contrast Sensitivity Between Measurements Immediately After Intervention and Measurements at Baseline
Description: Difference in contrast sensitivity was measured with the Pelli-Robson test, using a chart with letters arranged in groups of three. The first group has unit contrast and each subsequent group has a lower contrast. Passing a group means to read correctly at least two of the three letters. A Pelli-Robson score of 2.0 indicates normal contrast sensitivity of 100 percent. Scores less than 2.0 signify poorer contrast sensitivity. Pelli-Robson contrast sensitivity score of less than 1.5 is consistent with visual impairment and a score of less than 1.0 represents visual disability.
Time Frame: From baseline to time immediately after intervention
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Unit on a scale | 0.009 (0.282) | 0.018 (0.224)

7. Secondary Outcome: The Difference in Contrast Sensitivity Between Measurements at 3 Months After Intervention and Measurements at Baseline
Description: as for outcome 6
Time Frame: From baseline to 3 months
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Unit on a scale | 0.084 (0.205) | -0.026 (0.324)

8. Secondary Outcome: The Difference in Contrast Sensitivity Between Measurements at 6 Months After Intervention and Measurements at Baseline
Description: as for outcome 6
Time Frame: From baseline to 6 months
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Unit on a scale | 0.028 (0.221) | 0.009 (0.373)

9. Secondary Outcome: The Difference in Color Vision Between Measurements Immediately After Intervention and Measurements at Baseline
Description: The difference in color vision after intervention in comparison to Baseline was assessed by the investigator as 'Changed from Normal to Pathologic', 'Finding unchanged', and 'Changed from Pathologic to Normal'.
Time Frame: From baseline to time immediately after intervention
Population: Full Analysis Set (FAS)
Measure: Number; unit: Participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Participants
  Changed from Normal to Pathologic | 1 | 0
  Finding unchanged | 15 | 13
  Changed from Pathologic to Normal | 0 | 4

10. Secondary Outcome: The Difference in Color Vision Between Measurements at 3 Months After Intervention and Measurements at Baseline
Description: as for outcome 9
Time Frame: From baseline to 3 months
Population: Full Analysis Set (FAS)
Measure: Number; unit: Participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Participants
  Changed from Normal to Pathologic | 1 | 0
  Finding unchanged | 13 | 14
  Changed from Pathologic to Normal | 2 | 3

11. Secondary Outcome: The Difference in Color Vision Between Measurements at 6 Months After Intervention and Measurements at Baseline
Description: as for outcome 9
Time Frame: From baseline to 6 months
Population: Full Analysis Set (FAS)
Measure: Number; unit: Participants
Arm/Group | Alprostadil | Placebo
Number analyzed (Participants) | 16 | 17
Participants
  Changed from Normal to Pathologic | 1 | 0
  Finding unchanged | 12 | 15
  Changed from Pathologic to Normal | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to 33 weeks from first dose of trial medication on Day 1 to the last Follow-up Visit.
Description: AEs refer to the Safety Set (SS). The SS includes all randomized subjects who completed Visit 16 or terminated prematurely and who received at least one dose of trial medication.
Arm/Group | Alprostadil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 6/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alprostadil (N=18) | Placebo (N=18)
Choroidal Neovascularisation (Eye disorders) | 0 (0) | 1 (1)
Visual Disturbance (Eye disorders) | 0 (0) | 1 (1)
Vitreous Opacities (Eye disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Blood Pressure decreased (Investigations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.